CLINICAL TRIAL: NCT05124366
Title: Propolis Extract, Nanovitamin C and Nanovitamin E on Desquamative Gingivitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Rosa María López-Pintor Muñoz, Dos, PhD, Associate Professor., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0005
Record Dates: First submitted 2021-10-16; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Desquamative Gingivitis
Keywords: desquamative gingivitis; lichen planus; propolis
MeSH Terms: conditions — Gingival Diseases; Lichen Planus | interventions — Dental Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Nanovitamin E, nanovitamin C and propolis extract gel
  Interventions: Procedure: dental prophylaxis + oral hygiene instructions
- Placebo (Placebo Comparator): Gel without nanovitamin E, nanovitamin C and propolis extract
  Interventions: Procedure: dental prophylaxis + oral hygiene instructions

INTERVENTIONS:
Procedure: dental prophylaxis + oral hygiene instructions — Follow up: 2 weeks and 4 weeks

SUMMARY:
Objective: To evaluate the effectiveness of a gel containing nanovitamin C, nanovitamin E and propolis extract compared to a placebo in the treatment of desquamative gingivitis (GD) in patients with mucocutaneous diseases with gingival involvement. The possible improvement in the quality of life of these patients after treatment will also be evaluated.

Study design: Double-blind, randomized controlled study.

Patients: GD patients are being selected from the Postgraduate 'Specialist in Oral Medicine' of the Faculty of Dentistry, Complutense University of Madrid.

Allocation: Patients are being randomly assigned to the study group (dental prophylaxis + oral hygiene instructions + use of propolis gel for 4 weeks) or to the placebo group (dental prophylaxis + oral hygiene instructions + use of placebo gel for 4 weeks ). Both the study gel and the placebo are being used for brushing their teeth and for application in areas with GD.

Variables: The severity of the GD will be collected according to the scale of Arduino et al. 2017 and the periodontal variables (plaque index, probing bleeding index and probing depth). Pain during treatment will be recorded using a 10 cm visual analog scale (VAS). The quality of life in relation to oral health will be recorded using the Oral Health Impact Profile-14 (OHIP-14) questionnaire. These variables will be collected on day 0, 2 and 4 weeks after using the study gel or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age.
2. Patients with a clinical and histological diagnosis of some mucocutaneous disease. Patients diagnosed with oral lichen planus will be selected according to the American Academy of Oral and Maxillofacial Pathology, pemphigus vulgaris and / or scarring pemphigoid according to the 2015 World Workshop on Oral Medicine.
3. Patients who present GD, that is, erythema, epithelial desquamation, atrophy, painful erosions or ulceration of the free and / or attached gingiva, which is not related to the local accumulation of plaque.

Exclusion Criteria:

1. Being in cancer treatment with head and neck radiotherapy, chemotherapy or immunotherapy.
2. Being diabetic.
3. Being on topical corticosteroid treatment in the previous 4 weeks or systemic treatment in the previous 8 weeks.
4. Those patients who do not present the anterosuperior sector (from canine to upper canine) or the anteroinferior sector (from canine to lower canine) will also be excluded.
5. Pregnant or breastfeeding.
6. Being a smoker.
7. Use of rinses for plaque control.
8. Being medicated with drugs associated with gingival enlargement such as cyclosporine, calcium channel blockers and phenytoin.
9. To have taken antibiotics and / or anti-inflammatories 3 months before the study.
10. Taking medications capable of producing lichenoid reactions.
11. Patients who do not want to sign the informed consent.
12. Patients with periodontitis according to the consensus criteria of Papapanou et al. 2018 or patients treated for unstable periodontal disease according to the classification of Chapple et al. 2017.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The severity of the GD will be collected according to the scale of Arduino et al. 2017 | Baseline
  The Scale collects a value for each sextant in vestibular and another value in lingual / palatal (12 in total, six times vestibular and six times lingual / palatal). The criteria for scoring are as follows: (0) no detectable gingival lesions present, (1) only white lesions, (2) mild erythema (<3mm from the gingival margins), (3) one or more blisters or erythema clinically obvious (> 3mm from the gingival margins), (4) erosion or ulcer. When there are different characteristics, the clinician should choose the highest index, so the total score can vary from 0 to 48. Higher results indicate a more serious clinical disease.
The severity of the GD will be collected according to the scale of Arduino et al. 2017 | 2 weeks
  The Scale collects a value for each sextant in vestibular and another value in lingual / palatal (12 in total, six times vestibular and six times lingual / palatal). The criteria for scoring are as follows: (0) no detectable gingival lesions present, (1) only white lesions, (2) mild erythema (<3mm from the gingival margins), (3) one or more blisters or erythema clinically obvious (> 3mm from the gingival margins), (4) erosion or ulcer. When there are different characteristics, the clinician should choose the highest index, so the total score can vary from 0 to 48. Higher results indicate a more serious clinical disease.
The severity of the GD will be collected according to the scale of Arduino et al. 2017 | 4 weeks
  The Scale collects a value for each sextant in vestibular and another value in lingual / palatal (12 in total, six times vestibular and six times lingual / palatal). The criteria for scoring are as follows: (0) no detectable gingival lesions present, (1) only white lesions, (2) mild erythema (<3mm from the gingival margins), (3) one or more blisters or erythema clinically obvious (> 3mm from the gingival margins), (4) erosion or ulcer. When there are different characteristics, the clinician should choose the highest index, so the total score can vary from 0 to 48. Higher results indicate a more serious clinical disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We will try to publish it as a scientific article

REFERENCES:
- [Derived] Gonzalez-Serrano J, Serrano J, Sanz M, Torres J, Hernandez G, Lopez-Pintor RM. Efficacy and safety of a bioadhesive gel containing propolis extract, nanovitamin C and nanovitamin E on desquamative gingivitis: a double-blind, randomized, clinical trial. Clin Oral Investig. 2023 Feb;27(2):879-888. doi: 10.1007/s00784-022-04653-0. Epub 2022 Jul 28. PMID 35900605